CLINICAL TRIAL: NCT03374553
Title: A Prospective, Open, Multicentre Clinical Trial Analysing the Effectiveness and Safety of MINIject 636 in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Brief Title: MINIject 636 in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISM05
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: 26 patients enrolled into first arm, when enrolment completed, an additional 26 patients enrolled into second arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINIject DO Integrated System CS636 (MINI DO636) (Experimental): MINIject 636 implant is used to reduce intra-ocular pressure in the eye through a minimally-invasive glaucoma surgical intervention.
  The intervention is to be performed as stand-alone surgery. In this arm the implant is placed using Dual Operator Delivery Tool (DODT).
  Interventions: Device: MINI DO636
- MINIject SO Integrated System CS636 (MINI SO636) (Experimental): MINIject 636 implant is used to reduce intra-ocular pressure in the eye through a minimally-invasive glaucoma surgical intervention.
  The intervention is to be performed as stand-alone surgery. In this arm the implant is placed using Single Operator Delivery Tool (SODT).
  Interventions: Device: MINI SO636

INTERVENTIONS:
Device: MINI DO636 — MINIject 636 is an integrated system comprising a minimally-invasive Glaucoma Drainage Implant CS636 and a Delivery Tool.
  The Delivery Tool is a single-use tool, designed for inserting the CS636 implant into the sub-scleral location through an ab-interno minimally-invasive approach.
  For MINIject 636, there are 2 types of Delivery Tools available to implant and position the CS636 implant.
  Both types of Delivery Tools are being studied in this amended study: Dual Operator Delivery Tool (DODT) and Single Operator Delivery Tool (SODT).
  DODT is used in the first arm (cohort 1 - MINI DO636), SODT is used in the second arm (cohort 2 - MINI SO636).
  Arms: MINIject DO Integrated System CS636 (MINI DO636)
Device: MINI SO636 — MINIject 636 is an integrated system comprising a minimally-invasive Glaucoma Drainage Implant CS636 and a Delivery Tool.
  The Delivery Tool is a single-use tool, designed for inserting the CS636 implant into the sub-scleral location through an ab-interno minimally-invasive approach.
  For MINIject 636, there are 2 types of Delivery Tools available to implant and position the CS636 implant.
  Both types of Delivery Tools are being studied in this amended study: Dual Operator Delivery Tool (DODT) and Single Operator Delivery Tool (SODT).
  DODT is used in the first arm (cohort 1 - MINI DO636), SODT is used in the second arm (cohort 2 - MINI SO636).
  Arms: MINIject SO Integrated System CS636 (MINI SO636)

SUMMARY:
The study will evaluate the efficacy and safety of MINIject 636 and IOP lowering effects with or without glaucoma medications. The procedure will be a stand-alone surgery. Overall, the patient will be asked to perform several examinations up to 24 months after surgery.

The primary efficacy objective of the present study is to show the IOP reduction under medication 6 months after surgery compared to medicated diurnal IOP at screening.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary open angle glaucoma during screening/baseline visit or earlier.
* Grade 3 (open, 20-35 degrees) or grade 4 (wide open, 35-45 degrees) according to Shaffer Angle Grading System.
* Glaucoma not adequately controlled

Exclusion Criteria:

* Diagnosis of glaucoma other than open angle glaucoma
* Grade 2, grade 1 and grade 0 according to Shaffer Angle Grading System.
* Neovascular glaucoma in the study eye
* Prior glaucoma surgery in the study eye
* Clinically significant corneal disease
* Patients with poor vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Reduction in medicated diurnal IOP | 6 months after surgery
  DODT/SODT arm will be evaluated separately

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR Medical
Locations (3):
- Clínica Oftalmológica del Caribe, Barranquilla, Colombia
- Maxivision Eye Hospital, Hyderabad, Telangana, India
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No